CLINICAL TRIAL: NCT07396493
Title: A Prospective, Single-arm Study Evaluating the Endothelialization Effect and Timeline of AnchorMan® Left Atrial Appendage Occluder in Non-valvular Atrial Fibrillation Patients at High Risk of Stroke
Acronym: AnchorMan-NVAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Zhoupu Hospital, Pudong New Area, Shanghai, China (Other); Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-PM-02; 25SF1902201 (Other Grant/Funding Number: Shanghai Science and Technology Commission)
Record Dates: First submitted 2026-01-19; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF); High Risk of Stroke
Keywords: Non-valvular atrial fibrillation (NVAF); high risk of stroke.; Left Atrial Appendage Occluder System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): AnchorMan® Left Atrial Appendage Occluder System Treatment
  Interventions: Procedure: Intra-operative application of LAAC

INTERVENTIONS:
Procedure: Intra-operative application of LAAC — Undergoing left atrial appendage occlusion device for followup observation of the time course of device surface with the.endotheliation.

SUMMARY:
This study aims to evaluate the endotheliation efficacy of the AnchorMane® Left Atrial Appendage Occluder in non-valvular atrial fibrillation patients at high stroke risk. It investigates the rate of complete endotheliation of the occluder at 6 months post-procedure using routine cardiac CTA, providing additional data for clinical application and further product development.

Study Size and Duration: This study plans to enrol1 306 patients. All participants will undergo follow up immediately after occluder implantation, prior to discharge or within 7 days post-procedure, at 1 month post-procedure, at 3 months post-procedure,and at 6 months post-procedure. The total study duration is projected to be 3 year.

The expected duration of participation for each participant is approximately 6 months.

DETAILED DESCRIPTION:
Endothelialization within the left atrial appendage represents a core biological process following transcatheter left atrial appendage closure (LAAC). Advances in this field directly influence the optimization of postoperative anticoagulation strategies and the control of device related thrombosis (DRT) risks.

This multicenter, prospective, single-arm study primarily investigates the endotheliation efficacy of the AnchorMane® Left Atrial Appendage Occlusion Device using cardiac CTA following left atrial appendage occlusion. It plans to enroll 306 non-valvular atrial fibrillation patients undergoing left atrial appendage occlusion device for followup observation of the time course of device surface with the.endotheliation.

The device used in this study is the approved AnchorMane® Left Atrial Appendage Occlusion System, which is routinely employed in clinical practice.

What is required of me if I participate in the study?

If you decide to participate in this study, you will be enrolled after signing the informed consent form with full understanding. Participation in this trial requires your cooperation with the study physician to complete the following examinations or procedures :

* Baseline Visit (within 7 days pre-op): Collection of routine medical history, demographic data, physical examination,vital signs, modified Rankin Scale (mRS) score (if applicable), CHA2DS2,-VASc score.HAS-BLED score, NYHA functional class, electrocardiogram (EcG), laboratory tests(complete blood count, urinalysis, blood chemistry, coagulation profile, blood/urine pregnancy testif indicated, serum inflammatory markers),transesophageal echocardiography(TEE), and transthoracic echocardiography (TTE).
* Baseline Visit (Intra-operative): Vital signs, serum inflammatory markers, left atrial angiography, surgical records, medication records. Collect and document endpoint events and other adverse events.
* Discharge/Post-op 7-day Visit: Collect vital signs, modified Rankin Scale (mRS)score (if applicable), NYHA functional class, transthoracic echocardiogram (TTE), and laboratory test results (complete blood count, urinalysis, blood biochemistry, coagulation function, serum inflammatory markers)Complete medication records and collect/record for routine clinical care.information on endpoint events and other adverse events.
* 1-month Follow-up (±7 days): Collect results from routine diagnostic procedures including cardiac ultrasound (if applicable), cardiac CTA (if applicable), and laboratory tests.Complete documentation of medication history, endpoint events, and other adverse event information.
* 3-month Follow-up (±15 days): Complete and collect your routine clinical vital signs, cardiac ultrasound (if applicable), cardiac CTA, and serum inflammatory marker test results.Complete medication records, endpoint event documentation, and other adverse event records.
* 6-month Follow-up (±30 days): Complete and collect results of routine clinical examinations including vital signs, cardiac ultrasound, cardiac CTA, and serum inflammatory markers. Complete medication records, endpoint event documentation, and other adverse event records.
* Note: Laboratory tests included in the study comprise: Complete blood count : Collect hemoglobin, red blood cell, white blood cell, and platelet counts; Urinalysis: Collect urine red blood cells, urine white blood cells, urine protein, and urine glucose levels. Blood Biochemistry: Preoperative testing for total cholesterol, triglycerides,LDL cholesterol, HDl cholesterol, Creatinine, BUN, fasting blood glucose, albumin, ALT,AST; Pre-discharge Creatinine, alanine aminotransferase (ALT)，aspartatetests: aminotransferase (AsT). Coagulation function tests: Prothrombin time (PT), Prothrombintime international normalized ratio (INR), Activated partial thromboplastin time (APTT),Thrombin time (TT). Approximately 3 ml of blood will be drawn for each blood test, and approximately 3 ml of urine will be collected for each urine test. Your blood and urine samples will be used solely for routine hospital analysis and will not be sent externally.Remaining samples will be destroyed according to standard hospital protocols. During the study, we will need to collect your imaging data. This data will undergo de-identification and will be used exclusively for this research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with non-valvular atrial fibrillation (NVAF).
2. High stroke risk: CHA2DS2-VASc score ≥ 2 (Male) or ≥ 3 (Female) AND meeting any of the following:

   1. Documented history of bleeding (> 6 months ago) or bleeding tendency (e.g., gingival, nasal, GI, urinary tract, cerebral hemorrhage).
   2. Intolerance or unwillingness to undergo long-term anticoagulation therapy.
   3. Recurrent stroke or embolic events despite standardized anticoagulation.
   4. Predicted high bleeding risk (HAS-BLED score ≥ 3).
   5. Status post-Left Atrial Appendage Electrical Isolation (LAAEI).
3. Subject or legal representative understands the study purpose, is willing to cooperate with surgery and follow-up, and has signed the written Informed Consent Form (ICF).

Exclusion Criteria:

1. Rheumatic heart disease, moderate-to-severe mitral stenosis/regurgitation, severe aortic valve disease, or severe LVOT obstruction (gradient > 40 mmHg).
2. Left ventricular ejection fraction (LVEF) < 30%.
3. Complex LAA anatomy unsuitable for LAAO implantation.
4. Pericardial effusion > 10mm.
5. Planned ablation or cardioversion post-procedure.
6. Intracardiac thrombus (including left/right atrium).
7. Myocardial infarction within the last 3 months.
8. History of ASD repair or PFO occluder implantation.
9. History of heart valve replacement (mechanical valve).
10. Heart transplant recipient.
11. New-onset ischemic stroke or TIA within the last 30 days.
12. Severe heart failure (NYHA Class IV).
13. Severe renal impairment: eGFR < 45 ml/min/1.73m² or on dialysis.
14. Hypersensitivity or contraindication to aspirin, clopidogrel, heparin, contrast media, or nitinol.
15. Pregnant or lactating women, or those planning pregnancy within one year.
16. Life expectancy < 12 months.
17. Unable to complete 2 months of anticoagulation or 6 months of DAPT for any reason.
18. Investigator's judgment of poor compliance or inability to complete the study requirements.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-02-08 (Estimated); Primary Completion 2027-06-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete endothelialization rate of the LAA occluder | 6 months post-procedure.
  The proportion of subjects whose cardiac CTA shows complete endothelialization of the LAAO at 6 months post-occlusion. Complete endothelialization is defined as LAA density < 100 HU or < 25% of left atrial (LA) density under cardiac CTA examination.

SECONDARY OUTCOMES:
Device success rate | immediate post-procedure
  The proportion of subjects who correctly deployed and implanted the device in the appropriate location
Clinical success rate | 6 months post-operation
  The proportion of patients who do not experience ischemic stroke, hemorrhagic stroke, systemic embolism, cardiovascular death, or death of unknown cause after occlusion.
Procedural success rate | 7 days post-operation or at discharge
  Successful left atrial appendage occlusion with no device-related complications at discharge or within 7 days post-operation (whichever comes first).
Incidence of stroke and transient ischemic attack (TIA) | 3 months post-operation, 6 months post-operation
  Stroke is defined as all strokes in the Valve Research Consortium (VARC-3), specifically including ischemic stroke, hemorrhagic stroke, and undetermined stroke.
Incidence of systemic embolism | 3 months post-operation, 6 months post-operation
  Embolism other than stroke, such as myocardial infarction, pulmonary embolism, renal infarction, splenic infarction, limb ischemia, mesenteric ischemia, etc.
Serious bleeding events | before discharge or 7 days post-operation, 3 months post-operation, 6 months post-operation
  Serious bleeding refers to bleeding events of types 3-5 as defined in the Bleeding Research Consortium (BARC)
All-cause mortality | before discharge or 7 days post-operation, 3 months post-operation, 6 months post-operation
  Refer to the definition in VARC-3, which refers to death from any cause, including cardiovascular and non-cardiovascular death.
Incidence of Device-Related Complications | 6 Months Post-Op
  Device-related complications include device embolism, device corrosion, clinically significant device-to-surrounding structure interference, device thrombosis, device breakage, device infection/endocarditis/pericarditis, device perforation/tear, device allergy-induced cardiac tamponade, pericardial effusion requiring intervention, occluder embolism, and cardiac perforation.
Occluder Performance | 6 Months Post-Op
  Cardiac CTA or transesophageal (or chest wall) echocardiography was used to evaluate the device, including displacement, dislodgement, mitral regurgitation, residual shunt, and device-related thrombosis. The incidence of these events was calculated.
Left atrial appendage occluder complete endothelialization rate | 3 months post-operation
  The proportion of subjects whose cardiac CTA shows complete endothelialization of the LAAO at 3 months post-occlusion. Complete endothelialization is defined as LAA density < 100 HU or < 25% of left atrial (LA) density under cardiac CTA examination.
Device-related thrombosis (DRT) incidence | 3 months post-operation, 6 months post-operation
  assessed using cardiac CTA. DRT appears as a low-density filling defect on the left atrial side of the device surface. A thicker (>3 mm) and more prominent low-density defect is considered a typical manifestation of DRT.
Residual Leak (PDL) Incidence | before discharge or 7 days post-operation, 3 months post-operation, 6 months post-operation
  Cardiac CTA was used for assessment. A residual left atrial appendage density ≥100 HU or ≥25% of the left atrial density indicated the presence of a PDL. If TEE was used for assessment, residual shunts were classified based on color jet width as: minimal (1 mm), mild (1-3 mm), or relatively significant (3 mm). Complete closure was defined as no residual shunt greater than 5 mm on TEE examination.
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 3 months post-operation, 6 months post-operation
  MACCE includes perioperative complications and long-term follow-up complications. Specifically:
  * Perioperative complications: death, cardiac tamponade, device embolism, stroke, severe bleeding, and vascular access complications;
  * Long-term follow-up complications: ischemic stroke, hemorrhagic stroke, thromboembolism, device-related thrombosis, severe bleeding, and death.

OTHER OUTCOMES:
Serum inflammatory markers | preoperative, 24 hours postoperative, 1 week postoperative/before discharge (whichever comes first), 1 month postoperative, 3 months postoperative, 6 months postoperative
  Serum inflammatory markers[18] mainly include high-sensitivity C-reactive protein (Hs-CRP), interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), platelet-derived growth factor (PDGF), transforming growth factor-β (TGF-β), vascular endothelial growth factor (VEGF), fibroblast growth factor (FGF), matrix metalloproteinase-9 (MMP-9), and von Willebrand factor (vWF).

IPD SHARING:
Plan to Share IPD: No